CLINICAL TRIAL: NCT05525403
Title: The Effects of Fatigue on Exercise-Induced Hypoalgesia During a Dynamic Resistance Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Florida (Other)
Responsible Party: Principal Investigator, Abigail Wilson, Assistant Professor, University of Central Florida
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2
Record Dates: First submitted 2022-08-22; First posted 2022-09-01 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low Fatigue Exercise (Experimental): Participants will complete a single leg knee extension exercise with weight until they report a fatigue level = 3/10 on the Borg Rating of Perceived Exertion. Participants will complete three sets.
  Interventions: Other: Knee Extension Exercise
- High Fatigue Exercise (Experimental): Participants will complete a single leg knee extension exercise with weight until they report a fatigue level = 8/10 on the Borg Rating of Perceived Exertion. Participants will complete three sets.
  Interventions: Other: Knee Extension Exercise
- Quiet Rest (Active Comparator): Participants will rest quietly for two minutes, three sets.
  Interventions: Other: Quiet Rest

INTERVENTIONS:
Other: Knee Extension Exercise — Participants will be seated in a Steel Flex machine with weight equal to 50% of their 1 repetition maximum added to the machine. Participants will extend the dominant knee until the assigned fatigue level.
  Arms: High Fatigue Exercise; Low Fatigue Exercise
Other: Quiet Rest — Participants will sit quietly for two minutes, three times.
  Arms: Quiet Rest

SUMMARY:
The primary purpose of this study is to compare immediate changes in pain sensitivity (pressure pain threshold) during quiet rest, low fatigue exercise, and high fatigue exercise.

DETAILED DESCRIPTION:
Participants will attend three sessions. Participants will fill out questionnaires, undergo pain sensitivity testing, and be randomly assigned to complete a high and low fatigue exercise on either the second or third session. During the exercise, participants will complete three sets of a single leg knee extension exercise with weight equivalent to 50% of their 1 repetition maximum until they report either a high or low fatigue level. Immediately before and after each set, the research team will examine immediate changes in sensitivity to pressure (pressure pain threshold).

ELIGIBILITY:
Inclusion Criteria:

* Pain-free
* 18-60 years old
* Participant can appropriately perform the knee extension exercise (assessed during screening)

Exclusion Criteria:

* Non-English speaking
* Regular use of prescription pain medications
* Current or history of chronic pain condition
* Currently taking blood-thinning medication
* Systemic medical condition known to affect sensation, such as uncontrolled diabetes or neurological conditions
* Any contraindication to the application of ice, such as: uncontrolled hypertension (blood pressure over 140/90 mmHg), cold urticaria, cryoglobulinemia, paroxysmal cold hemoglobinuria, circulatory compromise
* Known presence of cardiovascular, pulmonary, or metabolic disease
* Current use of tobacco products
* Not physically ready to exercise without a medical exam as indicated by the Physical Activity Readiness Questionnaire Plus (PAR-Q+)
* Surgery, injury, or fracture to the lower back or lower extremity within the past 6 months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2022-10-28 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-04-20 (Actual)

PRIMARY OUTCOMES:
Change in Pressure Pain Threshold | Change from baseline immediately after exercise
  A digital pressure algometer will be applied to the quadriceps and upper trapezius for two trials each. Participants are instructed to say "stop" or "pain" so the stimulus can be terminated "when the sensation first transitions from pressure to pain" (pain threshold). Participants will rate the pain experienced during the threshold testing using a 101-point numeric pain rate scale (NPRS) anchored with 0= no pain to 100= the most intense pain sensation imaginable immediately following each testing time.

SECONDARY OUTCOMES:
Temporal Summation | Baseline, pre exercise
  Participants will rate a train of 10 heat pulses using the 101-point numerical pain rating scale
Heat Pain Threshold | Baseline, pre exercise
  A thermode will gradually increase temperature. Participants will state when the sensation first becomes painful.
Conditioned Pain Modulation | Baseline, pre exercise
  Pressure pain threshold after an ice water immersion task will be measured.
International Physical Activity Questionnaire Short Form | Baseline, pre exercise
  This is a self-report measure of physical activity that provides data regarding health-related physical activity.
Pittsburgh Sleep Quality Index | Baseline, pre exercise
  This is a 10-item questionnaire in which individuals respond to statements regarding sleep quality. A higher score indicates a worse sleep quality.
Pain Catastrophizing Scale | Baseline, pre exercise
  This is a 13-item questionnaire in which individuals respond to a statement on a five point scale from 0 to 4. Higher scores indicate higher pain catastrophizing levels.
Fear of Pain Questionnaire 9 | Baseline, pre exercise
  This is a 9-item questionnaire in which individuals respond to a statement on a five point scale from 1 to 5. Higher scores indicate higher fear of pain.
Pain Anxiety Symptom Scale | Baseline, pre exercise
  This is a 20-item questionnaire in which individuals respond to a statement on a six point scale from 0 to 5. Higher scores indicate higher pain-related anxiety.
Brief Resilience Scale | Baseline, pre exercise
  This is a 6-item questionnaire in which individuals respond to a statement on a five point scale from 1 to 5. Higher scores indicate greater resilience.
Preference for and Tolerance of the Intensity of Exercise Questionnaire | Baseline, pre exercise
  This is a 16-item questionnaire in which individuals respond to a statement on a five point scale from 1 to 5. Higher scores indicate lower tolerance for the intensity of exercise.

OTHER OUTCOMES:
1-repetition maximum testing | Baseline, pre exercise
  The amount of weight that can be lifted for 1 repetition

CONTACTS AND LOCATIONS:
Overall Officials: Abigail Wilson, Principal Investigator — University of Central Florida
Locations (1):
- University of Central Florida, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No